CLINICAL TRIAL: NCT06198387
Title: Efficacy and Safety of Radiotherapy for Prostate and Oligo-metastatic Lesions in Patients With Low-burden Oligo-metastatic Prostate Cancer: An Open, Exploratory Pilot Clinical Trial
Brief Title: Radiotherapy for Prostate and Oligo-metastatic Lesions in Patients With Low-burden Oligo-metastatic Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Changhai Hosp omPCa
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Oligo-metastatic Prostate Carcinoma
MeSH Terms: interventions — Hormones; abiraterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hormone and RT (Experimental): Patients with de novo oligo-metastatic prostate cancer will receive a two-year course of androgen deprivation therapy (ADT) in combination with abiraterone, along with synchronous metastasis-directed radiation and prostate radiotherapy.
  Interventions: Radiation: hormone and RT; Drug: ADT combined with abiraterone

INTERVENTIONS:
Radiation: hormone and RT — The patients will receive a two-year course of androgen deprivation therapy (ADT) in combination with abiraterone, along with synchronous metastasis-directed radiation and prostate radiotherapy(RT).
Drug: ADT combined with abiraterone — The patients will receive a two-year course of ADT combined with abiraterone.

SUMMARY:
The existing large prospective study demonstrates the benefits of primary radiotherapy in patients with low-volume oligo-metastatic prostate cancer (OMPC), and there is also more evidence of the benefits of local metastasis-directed therapy (MDT) for metastatic lesions. But there is no results from prospective study to demonstrate the efficacy of radiotherapy for prostate and oligo-metastases. Therefore, the aim of the protocol is to illustrate the efficacy of radiotherapy for prostate and oligo-metastatic lesions in patients with de novo OMPC.

DETAILED DESCRIPTION:
This study involves a single-center, limited-sample, single-arm exploration of radiotherapy for prostate and oligo-metastatic lesions in patients diagnosed with low-volume, hormone-sensitive OMPC. Eligible participants undergo thorough assessments and treatment involving endocrine therapy alongside radiation targeting metastatic lesions and the pelvic region. All patients received radiation therapy for both the primary and metastatic lesions combined endocrine therapy. Endocrine therapy with an antiandrogen (bicalutamide,for 4 weeks) androgen deprivation therapy combined with novel hormonal agents (acetate abiraterone), which will be continued for 2 years. The primary objective is to evaluate progression-free survival-2 (PFS-2), while secondary endpoints include ADT free survival, quality of life (QoL), overall survival, time to castration-resistant prostate cancer (CRPC), radiation-related complications and endocrine therapy related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over at the time of registration
* Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2;
* Histologically confirmed prostate adenocarcinoma via prostate biopsy;
* Assessment conducted via single-photon emission computed tomography (SPECT), magnetic resonance imaging (MRI), and Ga-68 prostate-specific membrane antigen (PSMA) positron emission tomography/computed tomography(PET/CT), revealing oligo-metastasis (involving < 4 metastatic lesions in non-pelvic lymph nodes and bones) with or without pelvic lymph node involvement;
* Expected survival duration >2 years.
* The willingness of patients to voluntarily accept the experimental research protocol after being informed of existing treatment options.

Exclusion Criteria:

* Any previous or ongoing treatment for prostate cancer, including radiotherapy, chemotherapy, focal treatment, etc.
* Pathology indicating small-cell or neuroendocrine tumor components;
* Patients with visceral metastases, or ≥4 metastases;
* Patients with concurrent malignancies or those in an acute infection period or severe infection state; patients positive for Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV), and/or syphilis (Treponema pallidum)
* Severe or active systemic comorbidities that, in the investigator's judgment, might interfere with the treatment, evaluation, and compliance of this trial, including severe conditions affecting respiratory, circulatory, nervous, mental, digestive, endocrine, immune, urological, and other systems;
* Individuals with contraindications related to radiation therapy may present heightened risks of treatment-related complications.
* Patients participating in other clinical trials;
* Patients unsuitable for participation in this clinical trial as per the judgement of the investigator.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival 2 (PFS2) | through study completion, an average of 3 years
  To assess the duration from the reinitiation of endocrine therapy until the identification of disease progression again.

SECONDARY OUTCOMES:
ADT free survival | through study completion, an average of 3 years
  To assess the timeframe between the completion of the initial ADT treatment and the onset of the subsequent ADT treatment.
self-assessment of quality of life (QoL) and patient satisfaction | through study completion, an average of 3 years
  To evaluate utilizing QoL questionnaires.In the EQ-5D descriptive system five dimensions are assessed: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Patients are asked to rate each dimension on a scale ranging from 'no problems'(1) to 'unable to/ extreme problems'(5).The VAS is a vertical scale ranging from 0 to 100 where 0 indicates worst imaginable health and 100 indicates best imaginable health.
5-year overall survival (OS) | Assessment overall survival (OS) at 5 years
  To assess the duration from enrollment until death from any cause or the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data including baseline characteristics,treatment information and follow-up data on toxicity, survival and disease control will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 5 years after the publication of the study.
Access Criteria: Data may be shared with radiation oncologists who are interested in examining the efficacy and toxicity of oligo-metastatic prostate cancer treated with radiation combined with drug or androgen deprivation therapy (ADT) combined with abiraterone. Detailed study protocol should be emailed along with the request of the data. The investigators may carefully review the study protocol, and data will only be shared with well-designed studies.

REFERENCES:
- [Derived] Xu B, Zhao X, Feng Z, Li J, Liang Y, Zhang W, Chen L, Shen X, Qu M, Gao X, Zhang H. Protocol for Evaluating the Efficacy and Safety of Radiotherapy for Prostate and Oligometastatic Lesions in Patients With Low-Burden Sensitive Oligometastatic Prostate Cancer: An Open, Exploratory Pilot Clinical Trial. Cancer Control. 2024 Jan-Dec;31:10732748241274595. doi: 10.1177/10732748241274595. PMID 39180187